CLINICAL TRIAL: NCT01324505
Title: An Open-label, One-sequence Cross-over, Single Centre Trial Investigating the Influence of Semaglutide on Pharmacokinetics of Ethinylestradiol and Levonorgestrel in an Oral Contraceptive Combination Drug After Multiple Dose Administration of Semaglutide in Subjects With Type 2 Diabetes
Brief Title: Effect of Oral Contraceptives After Administration of Semaglutide in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-3819; U1111-1119-2214 (Other: WHO); 2010-022435-11 (EudraCT Number)
Record Dates: First submitted 2011-03-25; First posted 2011-03-29 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One-sequence cross-over arm (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo; Drug: Microgyn®

INTERVENTIONS:
Drug: semaglutide — Semaglutide will be administered once weekly by s.c. (under the skin) injections in the abdomen. A total of 13 doses of semaglutide will be administered according to a predefined dosing scheme
Drug: placebo — Placebo semaglutide will be administered once for securing eligibility of subjects (willingness and ability to self inject) at the screening visit.
Drug: Microgyn® — Microgyn® will be given as once daily oral dosing in two periods, each of 8 days' duration. One tablet contains levonorgestrel 0.15 mg and ethinylestradiol 0.03 mg.

SUMMARY:
This clinical trial is conducted in Europe. The purpose of the trial is to investigate the influence on the pharmacokinetics (the rate at which the trial drug is eliminated from the body) of an oral contraceptive combination drug after multiple administration of semaglutide in female subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained by a physician before any trial-related activities
* Postmenopausal women: a. With at least 12 months of spontaneous amenorrhoea with serum follicle stimulating hormone (FSH) above 40 mIU/mL and oestrogen deficiency (estradiol levels less than 30 pg/mL, or a negative gestagen test) or b. Bilateral oophorectomy (surgical removal of both ovaries)
* Type 2 diabetes treated with either diet and exercise alone or with metformin (monotherapy) having a glycosylated haemoglobin (HbA1c) of 6.5 -10% (both inclusive)
* Stable treatment of diabetes, either diet and exercise only or a stable dose level of metformin, for at least 3 months
* BMI (Body Mass Index) between 18.5 - 35.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products
* Previous participation in this trial. Participation is defined as being dosed with either drug
* Treatment with antidiabetic drug other than metformin within the last 3 months
* Use of hormone replacement therapy within 4 weeks prior to starting dosing with the trial product
* Presence or history of cancer or any clinically significant diseases or disorders, considered by the physician to have influence on the results of this trial
* Subjects who are known to have hepatitis
* Positive human immunodeficiency virus (HIV) antibodies
* Uncontrolled treated/untreated hypertension (systolic blood pressure above 160 mmHg and/or diastolic blood pressure above 100 mmHg)
* History of alcoholism or drug abuse during the last 3 months
* History of chronic or idiopathic acute pancreatitis
* Family or personal history of multiple endocrine neoplasia type 2 (MEN2), or family history of medullary thyroid cancer (FMTC)
* Personal history of non-familial medullary thyroid carcinoma
* Subjects who are considered at increased risk of thrombosis formation, such as deep vein thrombosis, pulmonary embolism, infarction or apoplexy (as judged by the trial physician) and subjects who are smokers
* Blood or plasma donation within the last 3 months prior to first dosing
* Participation in any other trial investigating other products or involving blood sampling within the last 3 months prior to first dosing
* Inability or unwillingness to perform self-injection (with placebo medium) at trial start

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Area under the ethinylestradiol concentration-time curve | in the 24 hour dosing interval
Area under the levonorgestrel concentration-time curve | in the 24 hour dosing interval

SECONDARY OUTCOMES:
Maximum oral contraceptive concentration | in the 24 hour dosing interval
Area under the semaglutide concentration-time curve | in the 24 hour dosing interval
Maximum semaglutide concentration | within the weekly dosing interval
Percentage of subjects experiencing adverse events | from week 1 to end of trial at maximum 23 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Kapitza C, Nosek L, Jensen L, Hartvig H, Jensen CB, Flint A. Semaglutide, a once-weekly human GLP-1 analogue, does not reduce the bioavailability of oral contraceptives in patients with type 2 diabetes. Diabetes 2014; 63 (suppl 1): A595-A631 (2383-PO)
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com